CLINICAL TRIAL: NCT04983108
Title: Utility of Liver and Splenic Stiffness in Predicting Esophageal Varices in Patients With Acute on Chronic Liver Failure- A Cross-Sectional Study
Brief Title: Utility of Liver and Splenic Stiffness in Predicting Esophageal Varices in Patients With Acute on Chronic Liver Failure
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-07
Record Dates: First submitted 2021-05-31; First posted 2021-07-30 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2023-04

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACLF: ACLF
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention. This is an observational Study
  Other Names: This is an observational Study

SUMMARY:
Monitoring and Assessment: Transient Elastography will be performed in morning hours using the FibroScan apparatus (Echosens), which consists of a 5-MHz ultrasound transducer probe mounted on the axis of a vibrator. The tip of the transducer (M-or XL probe) will be covered with a drop of gel and placed perpendicularly in the intercostal space, with the patient lying in dorsal decubitus position with the right arm in the maximal abduction. Under control, in time motion and in A-mode, the operator will choose a liver portion within the right liver lobe, at least 6-cm thick and free of large vascular structures, and the gallbladder. Liver stiffness (LS) will be measured on a cylinder of hepatic tissue of 1 cm of diameter and 4 cm of length. For assessing the splenic stiffness (SS), the patient will be in supine position with left arm in maximum abduction. Ultrasonography will be used to identify and locate the spleen parenchyma, to choose the right place for SS measurement, and to measure the spleen diameter (long axis). Transducer will be placed in the left intercostal spaces, with location indicated by the ultrasound. A median value of 10 successful acquisitions, expressed in kPa, will be kept as a representative of the LS and SS measurements. The LS and SS measurement failure will be recorded when no value will be obtained after at least 10 shots. The results will be considered unreliable in the following circumstances: valid shots fewer than 10, success rate < 60%, or interquartile range / LS >30 %. Liver and splenic stiffness, LSPS score (LS measurement × spleen diameter / platelet count), Platelet count to spleen diameter ratio (PSR) will be calculated. Patient will also undergo upper g.i. endoscopy on same day. HVPG and TJLB will be done if indicated. The study will assess whether the stiffness scores correlate with presence of esophageal varices. Optimum cutoffs will be calculated for predicting the presence of esophageal varices.

* Study design: A Cross-Sectional Study
* Study period: 12 months
* Sample size with justification: Consecutive Patients of ACLF from approval of study to 12 months. ACLF patients will be screened and eligible patients will be taken in to the study.
* Intervention: Patients of ACLF will undergo upper g.i. endoscopy, liver and splenic stiffness measurement. HVPG and TJLB will be done in the patients only if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

- Patients of ACLF (APASL criteria).

Exclusion Criteria:

1. Age < 18 and > 70 years
2. moderate to severe ascites
3. Portal Vein Thrombosis
4. Hepatocellular carcinoma
5. space occupying lesion liver
6. heart failure
7. biliary obstruction
8. prior variceal endotherapy or ongoing beta blocker treatment for varices
9. pregnancy
10. ICD / pacemaker
11. ongoing treatment for HBV
12. HCV or ended within 3 months
13. No consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients of ACLF fulfilling the APASL (Asian Pacific Association for the Study of the Liver) criteria.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To assess the utility of liver and splenic stiffness and develop a model to predict presence of esophageal varices needing treatment in patients of ACLF. | Day 1

SECONDARY OUTCOMES:
To study the correlation of liver and splenic stiffness with grade of esophageal varices. | Day 1
To study utility of liver and splenic stiffness in evaluating esophageal varices in comparison with other non-invasive tests. | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided